CLINICAL TRIAL: NCT02109185
Title: A Randomized, Double-Blind, Multiple-Dose Trial of Mometasone Nasal Spray, 50 μg (Mylan), Nasonex® Nasal Spray, 50 μg (MSD-US), Nasonex® Nasal Spray Suspension, 50 μg (MSD-EU) & Placebo for Treatment of the Signs & Symptoms of Seasonal Allergic Rhinitis in 1,520 Male & Female Volunteers
Brief Title: A Comparison of Mometasone Nasal Spray, Nasonex Nasal Spray, Nasonex Nasal Spray Suspension, & Placebo for Treatment of Seasonal Allergies for Safety, Efficacy, & Superiority in 1520 Male & Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Organization: MylanPharma (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MOMT-12084
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Treatment of the Signs and Symptoms of Seasonal Allergic Rhinitis
Keywords: seasonal allergic rhinitis; grass/tree/ragweed allergies; nasal congestion/stuffiness; rhinnorea; nasal itching; sneezing
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Nasal Obstruction; Sneezing | interventions — alpha 1-Antichymotrypsin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mometasone Furoate Monohydrate Nasal Spray,50 μg/act. (Active Comparator): Days 1 through 7, each subject received a placebo run-in. Days 8 through 21, 2 sprays (2 × 50 μg) of Mometasone Furoate Monohydrate Nasal Spray per nostril once daily for 14 days. Total Daily Dose = 4 × 50 μg = 200 μg.
  Interventions: Drug: Mometasone Furoate Monohydrate Nasal Spray, 50 μg/act.
- Nasonex® Nasal Spray, 50 μg/actuation (Active Comparator): Days 1 through 7, each subject received a placebo run-in. Days 8 through 21, 2 sprays (2 × 50 μg) of Nasonex® Nasal Spray per nostril once daily for 14 days, Total Daily Dose = 4 × 50 μg = 200 μg.
  Interventions: Drug: Nasonex® Nasal Spray, 50 μg/actuation
- Nasonex® Nasal Spray Suspnsn, 50 μg/actuation (Active Comparator): Days 1 through 7, each subject received a placebo run-in. Days 8 through 21, 2 sprays (2 × 50 μg) of Nasonex® Nasal Spray Suspension per nostril once daily for 14 days, Total Daily Dose = 4 × 50 μg = 200 μg.
  Interventions: Drug: Nasonex® Nasal Spray Suspnsn, 50 μg/actuation
- Placebo Nasal Spray, 50 μL/actuation (Placebo Comparator): Days 1 through 7, each subject received a placebo run-in. Days 8 through 21, 2 sprays of placebo nasal spray per nostril once daily.
  Interventions: Drug: Placebo Nasal Spray, 50 μL/actuation

INTERVENTIONS:
Drug: Mometasone Furoate Monohydrate Nasal Spray, 50 μg/act.
  Arms: Mometasone Furoate Monohydrate Nasal Spray,50 μg/act.
Drug: Nasonex® Nasal Spray, 50 μg/actuation
  Arms: Nasonex® Nasal Spray, 50 μg/actuation
Drug: Nasonex® Nasal Spray Suspnsn, 50 μg/actuation
  Arms: Nasonex® Nasal Spray Suspnsn, 50 μg/actuation
Drug: Placebo Nasal Spray, 50 μL/actuation
  Arms: Placebo Nasal Spray, 50 μL/actuation

SUMMARY:
The study will compare the safety and efficacy of a generic mometasone nasal spray to the reference listed drugs in the treatment of seasonal allergic rhinitis. Additionally both the test and the reference formulations will be tested for superiority against a placebo nasal spray.

DETAILED DESCRIPTION:
The study is to compare the safety, efficacy, and superiority of generic mometasone nasal spray to reference products and to placebo in the treatment of seasonal allergic rhinitis. This protocol describes randomized, double-blind, placebo-controlled, 4- treatment group parallel study of 14 days duration preceded by a single blind 7-day placebo run-in period to investigate the clinical equivalence of Mylan's Mometasone Furoate Monohydrate Nasal Spray, 50 ug per actuation to Merck Sharp & Dohme's (MSD) Nasonex® Nasal Spray, 50 ug per actuation or MSD EU's Nasonex® Nasal Spray Suspension, 50 ug per actuation. In addition, the superiority of the test and reference products to placebo will be assessed. Prior to randomization to one of 4 study groups, each subject will have a 7-day placebo run-in period. Each subject will then receive one of the following treatments: Mylan's Mometasone Furoate Nasal Spray 50 μg/actuation (2 actuations per nostril per day); Merck-US Nasonex® Nasal Spray 50 μg/actuation (2 actuations per nostril per day); Merck-EU's Nasonex® and Nasal Spray Suspension 50 μg/actuation (2 actuations per nostril per day); or Mylan's Placebo Nasal Spray 50 μL/actuation (2 actuations per nostril per day). Active treatment is for 14 days duration. Reflective total nasal scores (rTNSS) will be collected every 12 hours for 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 12 years of age or older.
2. Signed informed consent form. For patients under the age of majority, the parent or legal guardian should sign the consent form and the child will be required to sign a patient "assent" form.
3. Sex: Male and/or non-pregnant, non-lactating females.

   * All women of childbearing potential must have a negative serum pregnancy test performed within 21 days prior to the start of the study and must be using a medically acceptable form of birth control.
   * Women will not be considered of childbearing potential if one of the following is reported and documented on the medical history:

     * postmenopausal with spontaneous amenorrhea for at least six months and a serum FSH levels >40mIU/ml, or
     * bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or
     * total hysterectomy and an absence of bleeding for at least 3 months.
4. History of seasonal allergic rhinitis of at least 2 years duration
5. Positive response to skin allergen testing to the relevant seasonal allergen (e.g. grass/tree/ragweed) for that sites geographical area within 14 months or at the time of study entry. Wheal size must be greater than or equal to (≥) 5 mm larger in diameter than diluent control via prick testing or greater than or equal to 7 mm larger in diameter than diluent control via intradermal testing.
6. Clinically active status (symptomatic) at both screening and baseline. The total nasal symptom score is to be greater than or equal to 6 on a 0-3 symptom scale with a score of at least 2 (moderate severity) for each of nasal congestion/stuffiness and one other nasal symptom score (rhinnorea, nasal itching, sneezing), and an overall disease rating of moderate or severe (e.g. total score of six or greater).
7. Weight: Age appropriate weight. BMI not to exceed 40 kg/m2
8. Tobacco Use: non-tobacco using for at least 3 months prior to study initiation.
9. Capable of providing informed consent or assent.
10. All subjects should be judged by the Principal Investigator or Medical Sub-Investigator as otherwise normal and healthy and free of clinically significant disease except for signs and symptoms of rhinoconjunctivitis that would interfere with the study schedule or evaluation of SAR during a pre-study medical evaluation performed within 21 days of the initial dose of study medication which will include:

<!-- -->

1. normal or non-clinically significant physical examination including nasal passage evaluation, including vital signs (pulse, temperature, respiration rate, blood pressure)
2. within normal limits or non-clinically significant laboratory evaluation results (unless otherwise specified) for the following tests:

   * Serum Chemistries
   * Sodium
   * Albumin
   * Blood urea nitrogen (BUN)
   * Potassium
   * Uric Acid
   * Aspartate aminotransferase (AST)
   * Chloride
   * Iron
   * Alanine aminotransferase (ALT)
   * Calcium *Total Cholesterol*
   * Alkaline Phosphatase
   * Creatinine *Glucose*
   * Phosphate
   * Total Protein *Triglycerides*
   * Total Bilirubin
   * Fasting or non-fasting may be performed based on clinical judgment

     - Hematology
   * Platelet Count
   * White blood cell count w/differential
   * Hemoglobin
   * Hematocrit
   * Red Blood Cell count

     * Urinalysis
   * Protein
   * pH
   * Specific Gravity
   * Appearance - Microscopic Examination (to be performed if urine dipstick is positive)
3. normal or non-clinically significant 12-lead ECG
4. negative urine drug screen including amphetamine, barbiturates, benzodiazepines, cannabinoid (marijuana), methadone, cocaine, opiates, and phencyclidine unless legal prescribed or allowed by state/federal law.
5. Additional tests and or examinations may be performed, if judged necessary by the Principal Investigator or Medical Sub-Investigator.

Exclusion Criteria:

1. Institutionalized subjects.
2. Individuals who have a rTNSS score of 6 or greater at the start of the placebo run-in period but who on the randomization day (i.e. Study Day 8) no longer meet the requirement (i.e. score <6) prior to randomization, or who have a score less than 2 for Stuffiness/Congestion, or who have a score of less than 2 for all 3 of the remaining Nasal Symptoms will result in discontinuation of the subject from the study and the subject will not receive randomized treatment. The rTNSS score assessed on the randomization day (i.e. Study Day 8) will be an average of the scores from the preceding 7 scoring time points. For example, if randomization occurs on Day 8, then the average total score of the placebo run-in phase will include the rTNSS scores from Study Day 5 (AM & PM), Study Day 6(AM & PM), Study Day 7(AM & PM), and Study Day 8(AM).
3. Females who are pregnant or nursing.
4. History of alcohol and/or drug abuse within 1 year of subject randomization.
5. Medications:

   *All routinely used (e.g. daily) concomitant medications taken for any co-morbidity (i.e. hypertension, high triglycerides, diabetes, etc) will be documented. Subjects receiving concomitant medications should be on stable doses of the medications (defined as no change in the dose for at least 3 months and the dose is not anticipated to change during the study).

   *Subject is dependent on nasal, oral, or ocular decongestants, or anti-inflammatory agents; as determined by the principal investigator, or diagnosis of rhinitis medicamentosa.

   *Subjects who cannot tolerate nasal sprays.

   *Use of intranasal or systemic first generation antihistamines, leukotriene receptor antagonists (i.e. montelukast) or other nasal decongestants within 3 days of enrollment.

   *Use of intranasal cromolyn within 14 days of enrollment.

   *Use of intranasal or systemic second-generation antihistamines (e.g. fexofenadine, loratadine, desloratadine, cetirizine) within 10 days of enrollment.

   *Use of any tricyclic anti-depressant within 30 days of enrollment.

   *Use of any ophthalmic steroids within 14 days or nasal, inhaled, or systemic steroids within 30 days of the study start. Super or high potency topical steroids should not be used during the study. The use of low potency topical corticosteroids will be allowed (e.g. over-the-counter 1% hydrocortisone).

   *Use of chronic medication that could affect the course of seasonal allergic rhinitis.
6. Diseases

   - Subjects who have had an upper respiratory tract or sinus infection requiring antibiotic therapy within thirty days days of enrollment, or who have had a viral upper respiratory tract infection within 30 days prior to the screening visit. History of recurrent sinusitis or chronic purulent postnasal drip

   - History of any significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychological, musculoskeletal disease, malignancies or other significant medical illness, which in the judgement of the principal investigator could interfere with the study or require medical treatment that would interfere with the study.

   - Clinical evidence of large nasal polyps, marked septal deviation, or any other nasal structural abnormality that may significantly interfere with nasal airflow, as determined by the principal investigator.
   * History of asthma over the previous two years that required chronic therapy with inhaled or systemic corticosteroids. Occasional acute or mild exercise induced asthma will be allowable on the condition that the treatment of the attacks is restricted to β-agonists only.
   * Recent exposure (within 30 days) or was at risk of being exposed to chicken pox or measles.
   * Previous seasonal allergic rhinitis or perennial allergic rhinitis that has proven unresponsive to steroid therapy.
   * Subjects with infectious rhinitis or atrophic rhinitis.
   * History of anaphylaxis and/or other severe local reactions(s) to skin testing, as determined by the Principal Investigator or Medical Sub-investigator.
   * Symptoms of common cold or upper respiratory infection or other acute illness at the screening or baseline visit.
   * Treatment for oral Candidiasis within 30 days of starting the study or a current oral Candidiasis infection
   * History of posterior subcapsular cataracts.
   * History of tuberculosis, or with the presence of uncontrolled glaucoma, cataracts, ocular herpes simplex, conjunctivitis or other eye infection not related to the diagnosis of seasonal allergic rhinitis.
   * Presence of untreated fungal, bacterial, or systemic viral infections within the previous 30 days.
7. Recent history of nasal septal surgery, nasal septal perforation (ulceration) or recent nasal injury that has not completely healed.
8. Any reason which, in the opinion of the Principal Investigator or Medical Sub-Investigator, would prevent the subject from safely participating in the study.
9. Travel outside the geographical region of pollen (local area) for more than 2 consecutive days or 3 days in total throughout the trial.
10. Anticipation of clinically significant symptoms due to perennial allergens (e.g. dust mite, molds, animal dander) prior to the anticipated start of the relevant seasonal allergy season. In other words anticipated flare of perennial allergy symptoms immediately prior to or during seasonal allergic rhinitis flare.
11. Previous participation in this study, or the patient is a member of the investigational study site staff or a member of the family of the investigational study site staff.
12. Not on stable dose of immunotherapy for at least 3 months prior to randomization and during trial.
13. Desensitization therapy to a seasonal allergen that is responsible for the subject's allergic rhinitis that is initiated or changed within the previous six months.
14. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
15. History of allergy/hypersensitivity to mometasone, other related products (i.e corticosteroids), or any of the inactive ingredients.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1307 (Actual)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Mean change from Baseline of the mean reflective Total Nasal Symptom Score (rTNSS) | 14 days
  The statistical analysis for both clinical equivalence and superiority of the active treatments over placebo will involve Analysis of Variance (ANOVA) and Analysis of Covariance (ANCOVA), respectively.
  The Per-Protocol Population (PPP) will be used for the primary analysis of bioequivalence.
  The Intent-to-Treat Population (ITT) will be used for the primary analysis of superiority.